CLINICAL TRIAL: NCT01542125
Title: The Effect of Liposomal Lidocaine on Perceived Pain in Children During Percutaneous Interosseous Pin Removal in the Outpatient Setting: A Triple Blinded, Randomized Placebo-controlled Clinical Trial
Brief Title: The Effect of Liposomal Lidocaine on Perceived Pain in Children During Percutaneous Interosseous Pin Removal in the Outpatient Setting
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RES0002737
Record Dates: First submitted 2011-12-15; First posted 2012-03-02 (Estimated); Results first posted 2016-05-23 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-06

CONDITIONS: Pain
Keywords: Patients aged 3 to 16 years presenting for; removal of smooth percutaneous interosseus pins; after orthopeadic surgery
MeSH Terms: conditions — Pain | interventions — Maxilene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Liposomal Lidocaine group (Experimental): Patients in this groups received 4% Liposomal Lidocaine that was applied to the area immediately surrounding the pin site(s) and was covered with an opaque Tegaderm dressing
  Interventions: Drug: Liposomal Lidocaine
- Placebo Group (Placebo Comparator): This group received a placebo that was applied to the area immediately surrounding the pin site(s) and was covered with an opaque Tegaderm dressing.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Liposomal Lidocaine — 4% Liposomal Lidocaine
  Other Names: Maxilene
  Arms: Liposomal Lidocaine group
Drug: Placebo — Tubes were visually identical to the Liposomal Lidocaine tubes.
  Arms: Placebo Group

SUMMARY:
The removal of smooth, percutaneous pins (Perc Pins), which are used for fracture fixation, occurs once adequate bone healing has taken place. At the Stollery Children's Hospital (SCH), this frequently performed procedure is currently done without anesthetic, making it a painful and uncomfortable experience for the child and their caregiver(s). Liposomal Lidocaine is a relatively new effective and "needle-free" topical anesthetic. The investigators were interested in examining its effectiveness in pain reduction in children undergoing Perc Pin removal. Objective: To determine if Liposomal Lidocaine is effective in reducing pain in a pediatric population undergoing Perc Pin removal compared to a placebo. Hypothesis: The investigators hypothesize that Liposomal Lidocaine would significantly reduce pain during Perc Pin removal compared to a placebo. Research Design: This was a triple-blinded, randomized placebo-controlled clinical trial with 281 patients (140 patients each in the Maxilene and 141 in the Placebo groups). Pain measurements, using the Oucher Scale (children) and a 10-cm Visual Analog Scale (parents and caregivers) were collected prior to randomization and immediately after Perc Pin removal. Data was analyzed using a Student's t-test and the Wilcoxon signed ranks test.

ELIGIBILITY:
Inclusion Criteria:

* Children between 3 and 16 years of age (i.e. up to but not including the 17th birthday) who present to the Pediatric Plaster Room at the SCH for Perc Pin removal were eligible for inclusion in this study.

Exclusion Criteria:

* Any patient with Perc Pins that are threaded (not smooth), as these pins require a more difficult removal process, oftentimes in the operating room instead of the orthopedic clinic.
* Infection around the Perc Pins: This is considered a relative contraindication to the use of topical anesthetic as it is usually less effective in this situation.
* Any parents/patients unable to exhibit understanding of the Oucher/VAS -- due to language barriers or developmental delay in the patient (e.g. severe cerebral palsy).
* The presence of an open wound in the vicinity of the pins that could not be excluded from the area to which the topical anesthetic cream is to be applied.
* Present use of analgesic or anxiolytic medications (within 24 hours prior to pin removal)
* Known allergies or adverse reactions to Maxilene

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 281 (Actual)
Dates: Start 2008-09; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sukhdeep Dulai, FRCSC, Principal Investigator — University of Alberta

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Liposomal Lidocaine Group | Placebo Group
Started | 140 | 141
Completed | 140 | 141
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Liposomal Lidocaine Group | Placebo Group | Total
Number analyzed (Participants) | 140 | 141 | 281
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.89 (3.71) | 7.74 (3.74) | 7.81 (3.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 63 | 123
  Male | 80 | 78 | 158

OUTCOME MEASURES:

1. Primary Outcome: Pain
Description: A horizontal 100 mm anchored Visual Analogue Scale (0 = no pain, 100 = worst possible pain) was used by the adult caregiver and the orthopedic technician to document the pain associated with Perc Pin removal for participant children.
  The Oucher Scale was used to assess pain intensity in participant children and included two separate scales. 6 photographs were assigned scores of 0, 20, 40, 60, 80, and 100 (in increasing increments of pain), such that these would be the scores averaged for participants unable to count by number. Children able to count to 100 by ones or tens and who could identify the larger of 2 numbers used the second scale; a vertical numeric one (0-100) that was printed next to the faces.
Time Frame: Before the application of Liposomal Lidocaine and immediately after Pin Perc removal, approximately 30 minutes
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Liposomal Lidocaine Group | Placebo Group
Number analyzed (Participants) | 140 | 141
units on a scale
  Pre-Pin Removal - Children, Oucher - Mean in mm | 0.70 (1.36) | 0.88 (1.9)
  Pre-Pin Removal - Parent, VAS - Mean in mm | 1.04 (1.63) | 0.87 (1.46)
  Pre-Pin Removal - Orthopedic Tec, VAS - Mean in mm | 0.27 (0.62) | 0.38 (0.92)
  Post-Pin Removal - Children, Oucher - Mean in mm | 3.03 (2.69) | 2.93 (2.94)
  Post-Pin Removal - Parent, VAS - Mean in mm | 3 (2.52) | 3.1 (2.60)
  Pos-Pin Removal - Orthopedic Tec, VAS - Mean in mm | 2.09 (1.93) | 2.06 (2.04)

ADVERSE EVENTS:
Arm/Group | Liposomal Lidocaine Group | Placebo Group
Serious Adverse Events (participants affected / at risk) | 0/140 | 0/141
Other Adverse Events (participants affected / at risk) | 0/140 | 0/141

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No